CLINICAL TRIAL: NCT03830463
Title: A Placebo-Controlled, Double-Blind, Single Ascending Dose Study to Evaluate the Safety and Pharmacokinetic Profile of CTP-692 in Fed and Fasted Conditions in Healthy Volunteers
Brief Title: Study to Assess the Safety and Pharmacokinetic (PK) of CTP-692 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP692.1002
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTP-692 (Experimental)
  Interventions: Drug: CTP-692
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTP-692 — Single oral dose
  Arms: CTP-692
Drug: Placebo — Single oral dose
  Arms: Placebo

SUMMARY:
This study will assess the safety and pharmacokinetic (PK) profile of single ascending doses of CTP-692 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 55 years of age, inclusive
* Body weight ≥ 55 kg and BMI within the range of 18 to 32 kg/m2, inclusive

Exclusion Criteria:

* Screening laboratory measurements outside the normal range associated with potential risk for the treatment under investigation at screening and/or prior to the first dose of study drug
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen or hepatitis C virus antibody
* History of clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal (GI) conditions
* Positive drug or alcohol test at screening or prior to the first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 48 hours
Measurement of CTP-692 exposure in plasma under fasted conditions | 48 hours
Measurement of CTP-692 exposure in plasma under fed conditions | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emily McIntyre, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No